CLINICAL TRIAL: NCT07002554
Title: The LIGHT-60 Trial - Light Intervention for Geriatric Patients Hospitalized for Depression Treatment
Brief Title: Bright Light Therapy for Depressed Geriatric Inpatients
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Benjamin Kalivas, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00139703; R25DA020537 (NIH)
Record Dates: First submitted 2025-05-06; First posted 2025-06-03 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Unipolar Depression
Keywords: Depression; Geriatrics; Psychiatry; Stress Disorders
MeSH Terms: conditions — Depressive Disorder; Depression; Stress Disorders, Traumatic | interventions — Ultraviolet Therapy; Phototherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright light therapy (Experimental): Participants in the intervention group will receive bright light therapy (BLT) consisting of 10,000 lux of bright white light administered for 30 minutes each morning, ideally within 30 minutes of awakening. Participants in both arms will continue to receive other treatment as usual (group therapy and medication management) as deemed appropriate by their treating clinicians.
  Interventions: Device: Bright light therapy
- Dim Red light (Sham Comparator): Participants in the control group will receive a placebo condition using an identical light box fitted with a translucent red screen to emit dim red light at an intensity of less than 2,500 lux, which lacks efficacy for depression treatment based on prior research. Participants in both arms will continue to receive other treatment as usual (group therapy and medication management) as deemed appropriate by their treating clinicians.
  Interventions: Device: dim red light

INTERVENTIONS:
Device: Bright light therapy — the Verilux® HappyLight® Lumi Plus light therapy box, which delivers UV-free, full-spectrum LED light at an intensity of 10,000 lux
  Other Names: light therapy
  Arms: Bright light therapy
Device: dim red light — The control group will use the same light box device, configured to emit dim red light. This will be achieved by setting the box to its lowest brightness setting and overlaying a translucent red filter over the light display. This setup is intended to maintain the appearance and experience of light exposure while minimizing any therapeutic effect.
  Arms: Dim Red light

SUMMARY:
Bright light therapy has been shown to be effective for the treatment of both seasonal and non-seasonal unipolar depression as well as bipolar depression, primarily in outpatients under the age of 60. There is a dearth of studies exploring the efficacy of this treatment modality among elderly depressed inpatients, which is our study population.

DETAILED DESCRIPTION:
Investigators are studying the ability of light therapy to reduce depressive symptoms in elderly patients who are hospitalized with unipolar depression (depression that is not due to bipolar disorder). Participants will receive either active light treatment or inactive treatment (also known as placebo).

ELIGIBILITY:
Inclusion criteria:

* A current episode of non-psychotic unipolar depression as the primary reason for psychiatric hospitalization
* Currently hospitalized on the MUSC Senior Care Unit
* Age 60 years or older
* HAMD-17 ≥8

Exclusion criteria:

* Any prior use of bright light therapy
* Primary indication for hospitalization is for a disorder other than major depressive disorder (determined by patient's treatment team)
* Photosensitive medical conditions or current use of photosensitizing medications - if patients have been advised by a treating clinician at any point to avoid sunlight because of their current medication regimen or medical condition, they will be considered to have a photosensitive medical condition and will be excluded from this study.
* Treatment with ECT; if a patient's condition deteriorates during study participation such that the treatment team feels ECT would be in their best interest, they will be withdrawn from study participation. For logistical and transport purposes, the study team feels that exclusion of patients receiving ECT will be necessarily. Additionally, these patients would likely be excluded from a future larger RCT given that ECT would likely interfere with signal of BLT efficacy.
* Uncontrolled headaches or any migraines within the last month
* Major neurocognitive disorder
* Severe intellectual disability
* Inability to consent for the study
* Active psychosis
* Inmates

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Study completion rate | Up to week 6 (Upon time of discharge from inpatient unit)
  Percentage of patients who complete the study while psychiatrically hospitalized
Adequacy of allocation blinding | Up to week 6 (Upon time of discharge from inpatient unit)
  assessed by the proportion of participants who correctly identify their study arm allocation. Blinding will be considered adequate if the proportion of correct guesses does not significantly exceed chance levels

SECONDARY OUTCOMES:
Preliminary efficacy data - Mean change in Hamilton Depression Rating Scale 17 item scale (HAMD-17) | Day of enrollment, week 1, week 2, week 4, week 6
  HAMD-17 is a commonly used clinician rating scale for depressive symptoms
Preliminary efficacy data - Mean change in Beck Depression Inventory II (BDI-II) Score | Day of enrollment, week 1, week 2, week 4, week 6
  BDI-II is a commonly used self-report rating scale for depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Rindy Fernandes, DO, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina Institute of Psychiatry Senior Care Unit, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao X, Ma J, Wu S, Chi I, Bai Z. Light therapy for older patients with non-seasonal depression: A systematic review and meta-analysis. J Affect Disord. 2018 May;232:291-299. doi: 10.1016/j.jad.2018.02.041. Epub 2018 Feb 17. PMID 29500957
- [Background] Geoffroy PA, Schroder CM, Reynaud E, Bourgin P. Efficacy of light therapy versus antidepressant drugs, and of the combination versus monotherapy, in major depressive episodes: A systematic review and meta-analysis. Sleep Med Rev. 2019 Dec;48:101213. doi: 10.1016/j.smrv.2019.101213. Epub 2019 Sep 18. PMID 31600678
- [Background] Oldham MA, Ciraulo DA. Bright light therapy for depression: a review of its effects on chronobiology and the autonomic nervous system. Chronobiol Int. 2014 Apr;31(3):305-19. doi: 10.3109/07420528.2013.833935. Epub 2014 Jan 7. PMID 24397276
- [Background] Tong H, Dong N, Lam CLM, Lee TMC. The effect of bright light therapy on major depressive disorder: A systematic review and meta-analysis of randomised controlled trials. Asian J Psychiatr. 2024 Sep;99:104149. doi: 10.1016/j.ajp.2024.104149. Epub 2024 Jul 15. PMID 39067131
- [Background] Menegaz de Almeida A, Aquino de Moraes FC, Cavalcanti Souza ME, Cavalcanti Orestes Cardoso JH, Tamashiro F, Miranda C, Fernandes L, Kreuz M, Alves Kelly F. Bright Light Therapy for Nonseasonal Depressive Disorders: A Systematic Review and Meta-Analysis. JAMA Psychiatry. 2025 Jan 1;82(1):38-46. doi: 10.1001/jamapsychiatry.2024.2871. PMID 39356500
- [Background] Sit DK, McGowan J, Wiltrout C, Diler RS, Dills JJ, Luther J, Yang A, Ciolino JD, Seltman H, Wisniewski SR, Terman M, Wisner KL. Adjunctive Bright Light Therapy for Bipolar Depression: A Randomized Double-Blind Placebo-Controlled Trial. Am J Psychiatry. 2018 Feb 1;175(2):131-139. doi: 10.1176/appi.ajp.2017.16101200. Epub 2017 Oct 3. PMID 28969438